CLINICAL TRIAL: NCT05031988
Title: Determinants of Physical Activity and Mental Health During and After Covid-19 Lockdown Among University Students
Brief Title: Determinants of Physical Activity and Mental Health During and After Covid-19 Lockdown
Status: Completed | Type: Observational
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Imtiyaz Ali Mir, Principal Investigator, Universiti Tunku Abdul Rahman
Other Study IDs: U/SERC/137/2021
Record Dates: First submitted 2021-09-01; First posted 2021-09-02 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: University Students

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- University Students: To assess the determinants of physical activity and mental health among university students during and after Covid-19 lockdown.
  Interventions: Other: No intervention will be used.

INTERVENTIONS:
Other: No intervention will be used. — Determinants of physical activity and mental health among the students during Covid-19 lockdown will be assessed.

SUMMARY:
Covid-19 pandemic has affected the entire globe for the past 2 years on a major scale, causing never before seen major effects on the way we live probably for the near future. SARS-Cov-2, previously known as coronavirus, is the causative virus for this disease and it originates from Wuhan, China with its first reported case of human infection back in December 2019. From there, it quickly resulted in an outbreak which was first unsuccessfully contained by the China government and has spread across the globe causing more than 187 million positive cases and 4.05 million deaths at the time of writing this proposal. For this reason, various measures have been implemented to control the spread of the virus with the main one to be discussed for reasons of this research, the movement restriction order (MCO). MCO was implemented to limit and control the local outbreak by restraining the movements of the people only to the absolute necessary. Social and religious gatherings, outdoor recreational activities, operation of learning institution of all levels are among those prohibited, only allowing essential goods store and health care facility centres to operate for the period.

Thus, this study is done to assess the impact Covid-19 movement restriction has had on university students from a physical and psychological standpoint during the MCO period. The implementation of the various restriction order has caused the students to go through numerous cycles of distress and it is of importance to determine the impact it has done to be able to provide the appropriate support if needed.

DETAILED DESCRIPTION:
Covid-19 by itself is a stressful and difficult health condition to face and deal with, as it not only affects people individually but threatens all those around them due to its highly contagious nature. As a public health emergency declared back in January 2020 by the WHO's Director, the primary worry for everyone is getting infected by the disease due to the ever increasing reported and suspected cases. This instils anxiety and fear and leads to all kinds of behaviours such as self-isolation, the worry of disseminating the disease to loved ones, and suspicion towards acquaintance that promotes paranoia and unhealthy thinking behaviours which propagate many psychological issues. Several studies on past pandemic have shown that these effects may extend to cause long term consequences on the relevant populations which is a concerning problem. Hawryluck et al. reported that following quarantine due to the SARS outbreak back in 2003, a substantial proportion of their participants still exhibits symptoms of Post-Traumatic Stress Disorder and depression. Bai et al study on health care workers during the same outbreak also reports quarantine being the most relevant factor for developing acute stress disorder and some of the participants considering resigning or being reluctant to work due to the outbreak. The health care workers were experiencing more exhaustion, restless sleep, and anxiety as well.

Tertiary level students consist of more out of state students, and this implies that most of them are probably living in hostels or near campus. The sudden lockdown that is imposed during June 2021 forced all the citizens to stay as they are, and prohibit socialization making a sudden change yet again to the environment university students are in after they could return to prepare for physical classes. This may induce a feeling of freedom being stripped away from university students, boredom when they are left all alone and uncertainty over their own health condition which all may prompt negative psychological impacts. The lockdown has also forced closure of academic institutions which leads to the teaching delivery to be converted from physical face-to-face to online. This can cause a whole lot of consequences. The primary concern for all the university students is definitely their academic progression. The students are now anxious about their study completion, whether they will be able to graduate on time and if their programme is still recognised. The running of the exams and those that are living with their family where they must share the load on household chores and taking care of their siblings or family members are some important stressors and can negatively affect thier mental health.

Maintaining PA has been well studied at this point for its effect on the physical health of an individual let it be better musculoskeletal health, reduced risk of developing cardiovascular diseases, or better self-esteem and confidence. Chekroud et al studied on the effect physical exercise has on mental health in their 1.2 million USA individuals and they report that generally physical activity has optimal effect on the mental health of their participants. Those who exercised have lower self-reported mental health burden than those who did not, and this association was consistent across all demographic factors be it age, gender, ethnicity, or household income. However, the type, duration, and intensity of exercise seems to have different ranges of response and it should be noted that more exercise is not always better. In their study, the duration of exercise between 30-60mins has the highest benefits in lowering mental health burden and this slowly declines with more duration of exercise and even worsen the mental state when it exceeds 3 hours.

To summarize, it is shown that physical activity is beneficial even for mental health and although the exact volume of physical exercise that's optimal is still up for discussion with further research delving into this area, we believe it is appropriate to say that exercise of any form is definitely better than being sedentary when it comes to the mental state of an individual. It is without a doubt a protective factor that everyone should maintain especially during these times of uncertainty to be in an optimal headspace. Therefore, aim of this study is to examine the determinanats of physical activity and mental health during and after Covid-19 lockdown among university Tunku Abdul Rahman students. Determinants of physcial activity and mental health are factors including gender, race, living condition, living area, restriction level, family income, and pre-lockdown habits that may or may not have effect on the differences in scores of the outcome measures.

Data will be tabulated into the microsoft excel, and analyzed with the help of SPSS (version 26). Mcnemer test will be used to compare the proportion of participans in each category (variables include gender, race, living condition, living area, restriction level, family income, and pre-lockdown habits) pre lockdown and post lockdown. Chi-square test would be utilized to assess if there is a significant difference between the groups (physically active vs inactive, anxiety vs no anxiety, depression vs no depression). Finally, logistic regeression will be implemented to determine the relationship of each variable with respect to outcome measures (physical activity, anxiety, and depression).

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students studying in Universiti Tunku Abdul Rahman, aged 18-25 years and are willing to participate in this study.

Exclusion Criteria:

* Students diagnosed with depression/anxiety or high stress before the implementation of movement control order.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy undergraduate students who are currently studying in Universiti Tunku Abdul Rahman without a previous history of depression, anxiety and/or stress.
Sampling Method: Non-Probability Sample
Enrollment: 442 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level | At baseline for a single time.
  Short form version of International Physical Activity Questionnaire (IPAQ-SF) will be used to determine the physical activity level of students. The questionnaire features 7 questions that relates to the frequency and duration the participant spends in various forms/intensity of physical activity over a period of one week and will categorize the participants into insufficiently active, minimally active and HEPA groups.
Depression | At baseline for a single time.
  Patient Health Questionaire-8 will be administered to evaluate the depression. Scoring of this questionnaire is based on a 4-point Likert scale, 0 having the least value and 3 maximum value.
Anxiety | At baseline for a single time.
  General Anxiety Disorder-7 scale will be used to examine the level of anxiety. Scoring of this questionnaire is based on a 4-point Likert scale, 0 having the least value and 3 maximum value.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Tunku Abdul Rahman, Kajang, Selangor, Malaysia